CLINICAL TRIAL: NCT03702283
Title: Effect of Providing Stratification of Low Risk Penicillin Allergies on Penicillin Allergy Label Removal in ICU Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Elizabeth J Phillips, Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 181734 -Pilot
Record Dates: First submitted 2018-10-08; First posted 2018-10-11 (Actual); Results first posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-01

CONDITIONS: Penicillin Allergy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Penicillin Allergic ICU Patients (Experimental): The intervention will provide access to a best-practices alert containing a penicillin allergy risk stratification tool and recommendations on whether to use an oral amoxicillin test dose challenge order set for patients who stratify as low risk.
  Interventions: Other: Penicillin Allergic Risk Stratification Best Practice Alert

INTERVENTIONS:
Other: Penicillin Allergic Risk Stratification Best Practice Alert — Providing best practice information on a patient's penicillin allergy risk and how to manage different levels of risk.

SUMMARY:
Currently it is estimated that at least 25 million people in the United States are labeled as penicillin allergic although less than 1.5 million of these are truly allergic. Although combined skin testing and oral challenge is an evidence-based de-labeling strategy the high burden of penicillin allergy labels means these services are available only through specialty allergy practices. There is therefore a need to provide evidence for alternative penicillin de-labeling strategies such as direct oral challenge. Previous studies have utilized quasi-experimental designs. Test dose challenges are currently recommended as a strategy for removal of low risk drug allergies, but the current experience is limited to single arm observational studies and evidence-based strategies for identifying low risk patients are lacking. The investigators objective is to demonstrate the benefit of providing risk stratification in removing penicillin allergy labels for low risk penicillin allergy patients in a single arm intervention pilot trial in the ICU setting, which will pave the way for a future stepped wedge randomized control trial (stepped wedge trial entered separately in clinical trials.gov as NCT03702270)

ELIGIBILITY:
Inclusion Criteria:

* VUMC patients age 18 or older with a penicillin allergy reported in their chart and are medically stable, currently admitted to ICU.

Exclusion Criteria:

* Patients with a penicillin allergy reported in their chart under ICU care, but who are currently medically unstable.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2019-03-31 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cosby A Stone, Jr., MD, Principal Investigator — Vanderbilt University Medical Center; Chris Lindsell, PhD, Study Chair — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Koo G, Stollings JL, Lindsell C, Dear ML, Kripalani S, Nelson GE, McCoy AB, Rice TW, Phillips EJ, Stone CA Jr; Vanderbilt University Medical Center Learning Healthcare System. Low-risk penicillin allergy delabeling through a direct oral challenge in immunocompromised and/or multiple drug allergy labeled patients in a critical care setting. J Allergy Clin Immunol Pract. 2022 Jun;10(6):1660-1663.e2. doi: 10.1016/j.jaip.2022.01.041. Epub 2022 Feb 5. No abstract available. PMID 35131513

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the two-year period from March 2019 to March 2021, a total of 5203 patients were admitted to the MICU, and 839 (16%) patients admitted to the MICU had a PAL. Of these, 240/839 (28.6%) of MICU patients with PALs met eligibility criteria and were determined to have low-risk PALs. Of those who were eligible, with a low-risk PAL, all 240 patients were offered an oral challenge with amoxicillin via informed consent, and 205/240 (85.4%) patients agreed to participate.
Pre-assignment Details: Of those who were eligible, with a low-risk PAL, all 240 patients were offered an oral challenge with amoxicillin via informed consent, and 205/240 (85.4%) patients agreed to participate.
Groups:
- Intervention Group- Single Arm: This study is a single arm intervention group study design in which patients with penicillin allergy labels (PALs) who were admitted to the Vanderbilt MICU were risk stratified into low-risk versus non-low risk penicillin allergies. Patients with low-risk penicillin allergies were offered the opportunity to receive a single dose 250mg amoxicillin challenge as a point of care test to remove their penicillin allergy at the point of care. Patients were potentially eligible for delabeling using amoxicillin challenge if they were hemodynamically stable, not pregnant, were cognitively capable of providing a history, (e.g. not delirious), and their PAL was low-risk.
Period: Overall Study
Arm/Group | Intervention Group- Single Arm
Started | 205 (Recruitment and observation began on March 31, 2019)
Completed | 205 (Recruitment and observation ended on March 31, 2021)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group- Single Arm: This study is a single arm intervention group study design in which patients with penicillin allergy labels (PALs) who were admitted to the Vanderbilt MICU were risk stratified into low-risk versus non-low risk penicillin allergies. Patients with low-risk penicillin allergies were offered the opportunity to receive a single dose 250mg amoxicillin challenge as a point of care test to remove their penicillin allergy at the point of care. Patients were potentially eligible for delabeling using amoxicillin challenge if they were hemodynamically stable, not pregnant, were cognitively capable of providing a history, (e.g. not delirious), and their PAL was low-risk.
  During the two-year period from March 2019 to March 2021, a total of 5203 patients were admitted to the MICU, and 839 (16%) patients admitted to the MICU had a PAL. Of these, 240/839 (28.6%) of MICU patients with PALs met eligibility criteria and were determined to have low-risk PALs. Of those who were eligible, with a low-risk PAL, all 240 patients were offered an oral challenge with amoxicillin, and 205/240 (85.4%) patients agreed.
Arm/Group | Intervention Group- Single Arm
Number analyzed (Participants) | 205
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [48 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 112
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 202
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 21
  White | 179
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 205

OUTCOME MEASURES:

1. Primary Outcome: Penicillin Allergy Label Removal
Description: The proportion of patients with low risk penicillin allergy whose labels are removed from the medical chart's allergy section.
Time Frame: Hospital discharge at approximately 7 days after ICU transfer
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group- Single Arm
Number analyzed (Participants) | 205
Participants | 201

2. Primary Outcome: Patients With Low Risk Penicillin Allergy Label Who Underwent Amoxicillin Challenge
Description: The proportion of patients with low risk penicillin allergy who underwent amoxicillin challenge
Time Frame: Hospital discharge at approximately 7 days after ICU transfer
Population: Baseline for this measure is those who were offered amoxicillin challenge, rather than those who agreed to it.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group- Single Arm
Number analyzed (Participants) | 240
Participants | 205

3. Secondary Outcome: Adverse Events (in Particular, Reported Allergic Events)
Description: The proportion of penicillin allergic patients challenged with amoxicillin who reported adverse events
Time Frame: Hospital discharge at approximately 7 days after ICU transfer
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group- Single Arm
Number analyzed (Participants) | 205
Participants | 1

4. Secondary Outcome: Communication About Penicillin Allergy in Discharge Summary
Description: The proportion of penicillin allergic patients whose discharge summary contains information about penicillin allergy at discharge.
Time Frame: Hospital discharge at approximately 7 days after ICU transfer
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group- Single Arm
Number analyzed (Participants) | 205
Participants | 202

5. Secondary Outcome: Antibiotic Utilization by Patients
Description: The number of changes or new starts of penicillin treatments as a result of penicillin allergy label removal and the proportion of patients experiencing this event
Time Frame: 2 years observation
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group- Single Arm
Number analyzed (Participants) | 205
Participants | 59

ADVERSE EVENTS:
Time Frame: For adverse events associated with challenge, 7 days of follow up were collected. For adverse events during subsequent penicillin treatments at VUMC, 2 years of follow up data were collected.
Arm/Group | Intervention Group- Single Arm
All-Cause Mortality (participants affected / at risk) | 0/205
Serious Adverse Events (participants affected / at risk) | 1/205
Other Adverse Events (participants affected / at risk) | 2/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group- Single Arm (N=205)
Morbilliform Exanthem following Amoxicillin Challenge (Skin and subcutaneous tissue disorders) | 1 (1) — Morbilliform Drug Exanthem
Morbilliform Exanthem During Subsequent Penicillin Treatment at VUMC (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group- Single Arm (N=205)
Gastrointestinal Intolerance During Subsequent Penicillin Treatment at VUMC (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT03702283/Prot_SAP_000.pdf